CLINICAL TRIAL: NCT00990158
Title: A Multicentre Study of Low Dose Oral Vitamin K for INR Control in Patients Receiving Warfarin
Brief Title: Does Low Dose Oral Vitamin K Improve International Normalized Ratio (INR) Stability?
Acronym: OVWAC VII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other); University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Mark Crowther, Vice President, Research, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA 6695
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2013-12

CONDITIONS: Coagulation; Bleeding; Thrombosis
Keywords: Vitamin K1 (phytonadione); Randomized controlled trial; Warfarin; Coagulopathy; Time in therapeutic range; Bleeding; Thrombosis; VKORC1 and CYP2C9 genotypes; Time INR in therapeutic range
MeSH Terms: conditions — Thrombosis; Hemorrhage; Hemostatic Disorders; Vitamin K-Dependent Clotting Factors, Combined Deficiency Of, Type 2 | interventions — Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose vitamin K + usual warfarin (Active Comparator): Low dose oral vitamin K (0.150 mg orally once daily) + warfarin continuation with usual warfarin monitoring
  Interventions: Drug: Phytonadione (Vitamin K1)
- Usual warfarin therapy + placebo (Placebo Comparator): Patients continue usual warfarin and take one placebo per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Phytonadione (Vitamin K1) — A daily dose of 150 micrograms of vitamin K medication given orally for a total of 7 months
  Arms: Low dose vitamin K + usual warfarin
Drug: Placebo — A daily dose of matching placebo medication given orally for a total of 7 months
  Arms: Usual warfarin therapy + placebo

SUMMARY:
Warfarin is highly effective for the prevention of both first and recurrent thrombotic events, however even minor excursions outside the reference INR range of 2.0 to 3.0 are associated with bleeding or thrombotic complications. The importance of maintaining the INR within the desired interval has led to the concept of "time in therapeutic range (TTR)" - the total proportion of time that the INR is between 2.0 and 3.0. The investigators propose a multicentre, double blind, randomized trial which will determine if 0.150 mg of oral vitamin K increases time in the therapeutic range for patients receiving warfarin.

DETAILED DESCRIPTION:
What is/are the principal research objective(s) and question(s) to be addressed? Research Objectives: Our broad objective is to improve the quality of anticoagulant care for patients receiving warfarin. Our specific objective is to determine if we can improve the TTR with LDVK, a non-toxic, inexpensive and easily administered medication.

Hypothesis: We hypothesize that patients receiving vitamin K will have a higher TTR than those receiving placebo. In a mechanistic study we proposed that VKORC1 and CYP2C9 genotype will modulate the impact of vitamin K on INR control.

Research questions:

Efficacy (primary): When compared with placebo does the addition of 150 micrograms of daily vitamin K to "usual warfarin therapy" improve anticoagulant control as measured by "time in the therapeutic range"? Safety (Secondary): Does LDVK increase the frequency of adverse clinical events, including thromboembolism? Does LDVK reduce the risk of major and/or all bleeding? Mechanistic (Hypothesis generating): Do VKORC1 and CYP2C9 genotypes modulate the effect vitamin K on INR stability?

Study design:

The proposed pilot study is a multi-centre, placebo controlled, randomized trial with an additional pilot mechanistic study (Figure 1 provides a broad outline of the study).

Study interventions:

Patients will receive a daily dose of 150 micrograms of vitamin K or a matching placebo medication for a total of 7 months - a one month "run in period" and a 6 month period of follow-up. They will continue to receive warfarin under the supervision of their anticoagulant clinic - other than one study mandated INR within 7 days of enrolment no changes in patient care will be made as a result of participation in this study.

All patients will be enrolled in a mechanistic study. Patients will have blood drawn at the time they provide consent to have their VKORC1 and CYP2C9 genotypes determined.

Allocation of patients into study groups:

Randomization will be achieved using a computer generated random number table. Patients will be stratified based on clinical centre. Practically, a random number table will be produced at the coordinating centre for each clinical centre. The study coordinating centre will package a six week supply of drug and placebo into sequentially numbered, identical drug containers based on the randomization sequence for each site. The drug packages will then be shipped to each centre. After consent is obtained, and the coordinating centre is notified, patients will be allocated to treatment by dispensing sequential drug containers in numeric sequence. Additional supplies (for a total of seven months of therapy for each patient) will be dispensed by the anticoagulant clinic in blocks of 6 weeks. This method of allocation ensures research subjects and study staff are masked to allocation as drug and placebo are identical. Masked allocation will be further protected by not providing an unblinding schedule for centres as we can foresee no circumstance in which immediate unblinding would be required.

Frequency and duration of trial follow-up:

Patients will have their INR checked at a minimum of 1 week after initiation of study drug and then will be followed as per their anticoagulant clinic routine. We will not mandate any particular frequency of INR testing as changing clinic routines will induce unwanted changes in INR control is a co-intervention that could influence TTR and that is not attributable to the study intervention. Clinical events will be reviewed, as per current clinic routine, at each INR check. If clinical events are reported source documentation will be sought for the purposes of adjudication. Our research group has extensive prior experience with collection and interpretation of INR values, and of the ascertainment, collection and reporting of clinical events in anticoagulated patients.

Primary and secondary outcome measures:

The primary outcome is a simple comparison of mean TTRs in the LDVK and placebo patients. As noted, calculation of the TTR will begin at the first INR obtained a minimum of 4 weeks after randomization and will end 7 months after enrolment. The TTR will be calculated using a previously validated computer algorithm, based on the method of Rosendaal et al (7). Secondary outcome measures will include (a) all significant INR excursion (INR < 1.5 or > 4.5), (b) number of INR determinations and (c) bleeding and thrombotic events of sufficient severity to require a medical intervention - where possible source documents from hospital admissions will be obtained to allow characterization of these events. Major bleeding will be defined as bleeding consistent with the 8th ACCP guidelines (36). All bleeding and thrombotic events will be independently adjudicated by a panel of experts based on submitted source documentation.

Plan for ascertaining outcome measures at follow-up:

INR values are obtained routinely as part of warfarin care. All INR determinations will be performed in clinical laboratories that participate in provincially mandated external quality assessment exercises to ensure quality. INR values and current warfarin dose will be reported to the coordinating centre using the online data entry and reporting system. Clinical events will be measured as per the "Primary and secondary outcome measures" section.

Will health services research issues be addressed within this trial? As a pilot study we do not feel that a valid health services research question can be posed in the context of this study. We do propose a simple cost effectiveness analysis which will examine the estimated total costs of participation in the study - for this analysis we will compare the number and type of medical interventions (and their costs) in the two arms of the study. Costs will be determined from validated Ontario costing data for INR tests, clinical visits and monitoring costs as well as any estimated costs attributable to clinic events, should these occur. Funding for this analysis will be sought from different sources, however we will ensure that the data required to complete this analysis will be collected within the context of this study.

Trial sample size and justification for the assumptions underlying the power calculations:

As a pilot study of a novel intervention we do not have estimates of the improvement of the TTR we expect to see with LDVK. As such the proposed sample size of 400 patients (200 per arm) is one of convenience however the study is powered to detect probable changes in TTR. Thus, we have an 85% likelihood of detecting a 15% increase in TTR assuming a TTR of 55% in the placebo arm (two sided alpha = 0.05, comparison of proportions, Fleiss correction) (37). A table of conditional powers is presented in Table 2. In subsequent studies (if justified, based on the results of this study) we will power based on the rates of clinical events. One prior paper has examined increases in TTR with vitamin K administration; the increase in TTR in this study was 28%, thus we are reassured by our ability to reliably detect a 15% difference in TTR (17).

ELIGIBILITY:
Inclusion Criteria:

* Warfarin therapy administered to a target INR of 2.0 to 3.0

Exclusion Criteria:

* Out of range INR on day of screening - enrolment will only occur if the patient's INR on the day of screening is between 1.8 and 3.4 (inclusive) - if the INR is outside this range the patient will be re-screened when the INR is within this range.
* Recent warfarin initiation - all patients must have received warfarin for a minimum of 3 months
* Planned termination or extended temporary interruption of warfarin within 6 months or anticipated survival of less than 6 months
* Known severe liver disease, known excess alcohol consumption , known malabsorption syndrome or inability to take oral medications
* Use of medications known to interfere with warfarin and whose dose is likely to change over the course of the study (e.g. barbiturates, rifampin etc.)
* Known allergy to vitamin K
* Inability or unwillingness to follow study procedures or provide consent
* Prior participation in this study, or participating in a competing study which may impact INR control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2010-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
When compared with placebo does the addition of 150 micrograms of daily vitamin K to "usual warfarin therapy" improve anticoagulant control as measured by "time in the therapeutic range"? | 7 Months

SECONDARY OUTCOMES:
Does low dose Vitamin K (LDVK) increase the frequency of adverse clinical events, including thromboembolism and major and/or all bleeding? | 7 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Crowther, MD, Principal Investigator — McMaster University
Locations (4):
- Canada (4):
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - University Health Network, Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Background] Ansell J, Hirsh J, Hylek E, Jacobson A, Crowther M, Palareti G. Pharmacology and management of the vitamin K antagonists: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):160S-198S. doi: 10.1378/chest.08-0670. PMID 18574265
- [Background] Oake N, Jennings A, Forster AJ, Fergusson D, Doucette S, van Walraven C. Anticoagulation intensity and outcomes among patients prescribed oral anticoagulant therapy: a systematic review and meta-analysis. CMAJ. 2008 Jul 29;179(3):235-44. doi: 10.1503/cmaj.080171. PMID 18663203
- [Background] Dentali F, Douketis JD, Lim W, Crowther M. Combined aspirin-oral anticoagulant therapy compared with oral anticoagulant therapy alone among patients at risk for cardiovascular disease: a meta-analysis of randomized trials. Arch Intern Med. 2007 Jan 22;167(2):117-24. doi: 10.1001/archinte.167.2.117. PMID 17242311
- [Background] Kaufman DW, Kelly JP, Rosenberg L, Anderson TE, Mitchell AA. Recent patterns of medication use in the ambulatory adult population of the United States: the Slone survey. JAMA. 2002 Jan 16;287(3):337-44. doi: 10.1001/jama.287.3.337. PMID 11790213
- [Background] Verhovsek M, Motlagh B, Crowther MA, Kennedy C, Dolovich L, Campbell G, Wang L, Papaioannou A. Quality of anticoagulation and use of warfarin-interacting medications in long-term care: a chart review. BMC Geriatr. 2008 Jul 3;8:13. doi: 10.1186/1471-2318-8-13. PMID 18598364
- [Background] Schmitt L, Speckman J, Ansell J. Quality assessment of anticoagulation dose management: comparative evaluation of measures of time-in-therapeutic range. J Thromb Thrombolysis. 2003 Jun;15(3):213-6. doi: 10.1023/B:THRO.0000011377.78585.63. PMID 14739631
- [Background] Rosendaal FR, Cannegieter SC, van der Meer FJ, Briet E. A method to determine the optimal intensity of oral anticoagulant therapy. Thromb Haemost. 1993 Mar 1;69(3):236-9. PMID 8470047
- [Background] Pirmohamed M, James S, Meakin S, Green C, Scott AK, Walley TJ, Farrar K, Park BK, Breckenridge AM. Adverse drug reactions as cause of admission to hospital: prospective analysis of 18 820 patients. BMJ. 2004 Jul 3;329(7456):15-9. doi: 10.1136/bmj.329.7456.15. PMID 15231615
- [Background] Wysowski DK, Nourjah P, Swartz L. Bleeding complications with warfarin use: a prevalent adverse effect resulting in regulatory action. Arch Intern Med. 2007 Jul 9;167(13):1414-9. doi: 10.1001/archinte.167.13.1414. PMID 17620536
- [Background] Sconce EA, Avery PJ, Wynne HA, Kamali F. Vitamin K epoxide reductase complex subunit 1 (VKORC1 ) polymorphism influences the anticoagulation response subsequent to vitamin K intake: a pilot study. J Thromb Haemost. 2008 Jul;6(7):1226-8. doi: 10.1111/j.1538-7836.2008.03003.x. Epub 2008 Jul 1. No abstract available. PMID 18466315
- [Background] Sconce E, Khan T, Mason J, Noble F, Wynne H, Kamali F. Patients with unstable control have a poorer dietary intake of vitamin K compared to patients with stable control of anticoagulation. Thromb Haemost. 2005 May;93(5):872-5. doi: 10.1160/TH04-12-0773. PMID 15886802
- [Background] Khan T, Wynne H, Wood P, Torrance A, Hankey C, Avery P, Kesteven P, Kamali F. Dietary vitamin K influences intra-individual variability in anticoagulant response to warfarin. Br J Haematol. 2004 Feb;124(3):348-54. doi: 10.1046/j.1365-2141.2003.04787.x. PMID 14717783
- [Background] Cushman M, Booth SL, Possidente CJ, Davidson KW, Sadowski JA, Bovill EG. The association of vitamin K status with warfarin sensitivity at the onset of treatment. Br J Haematol. 2001 Mar;112(3):572-7. doi: 10.1046/j.1365-2141.2001.02635.x. PMID 11260056
- [Background] Reese AM, Farnett LE, Lyons RM, Patel B, Morgan L, Bussey HI. Low-dose vitamin K to augment anticoagulation control. Pharmacotherapy. 2005 Dec;25(12):1746-51. doi: 10.1592/phco.2005.25.12.1746. PMID 16305294
- [Background] Booth SL, Charnley JM, Sadowski JA, Saltzman E, Bovill EG, Cushman M. Dietary vitamin K1 and stability of oral anticoagulation: proposal of a diet with constant vitamin K1 content. Thromb Haemost. 1997 Mar;77(3):504-9. PMID 9066002
- [Background] Bovill EG, Fung M, Cushman M. Vitamin K and oral anticoagulation: thought for food. Am J Med. 2004 May 15;116(10):711-3. doi: 10.1016/j.amjmed.2004.02.020. No abstract available. PMID 15121498
- [Background] Sconce E, Avery P, Wynne H, Kamali F. Vitamin K supplementation can improve stability of anticoagulation for patients with unexplained variability in response to warfarin. Blood. 2007 Mar 15;109(6):2419-23. doi: 10.1182/blood-2006-09-049262. Epub 2006 Nov 16. PMID 17110451
- [Background] Rombouts EK, Rosendaal FR, Van Der Meer FJ. Daily vitamin K supplementation improves anticoagulant stability. J Thromb Haemost. 2007 Oct;5(10):2043-8. doi: 10.1111/j.1538-7836.2007.02715.x. Epub 2007 Jul 31. PMID 17666020
- [Background] de Assis MC, Rabelo ER, Avila CW, Polanczyk CA, Rohde LE. Improved oral anticoagulation after a dietary vitamin k-guided strategy: a randomized controlled trial. Circulation. 2009 Sep 22;120(12):1115-22, 3 p following 1122. doi: 10.1161/CIRCULATIONAHA.109.849208. Epub 2009 Sep 8. PMID 19738137
- [Background] Schurgers LJ, Shearer MJ, Hamulyak K, Stocklin E, Vermeer C. Effect of vitamin K intake on the stability of oral anticoagulant treatment: dose-response relationships in healthy subjects. Blood. 2004 Nov 1;104(9):2682-9. doi: 10.1182/blood-2004-04-1525. Epub 2004 Jul 1. PMID 15231565
- [Background] Ford SK, Misita CP, Shilliday BB, Malone RM, Moore CG, Moll S. Prospective study of supplemental vitamin K therapy in patients on oral anticoagulants with unstable international normalized ratios. J Thromb Thrombolysis. 2007 Aug;24(1):23-7. doi: 10.1007/s11239-007-0014-z. Epub 2007 Feb 24. PMID 17323135
- [Background] Crowther MA, Ageno W, Garcia D, Wang L, Witt DM, Clark NP, et al. Effectiveness of low dose oral vitamin K for patients with elevated INR values: results of a randomized trial examining clinical outcomes. Journal of Thrombosis & Haemostasis 5[S2], PS 219. 2008.
- [Background] Woods K, Douketis JD, Kathirgamanathan K, Yi Q, Crowther MA. Low-dose oral vitamin K to normalize the international normalized ratio prior to surgery in patients who require temporary interruption of warfarin. J Thromb Thrombolysis. 2007 Oct;24(2):93-7. doi: 10.1007/s11239-007-0022-z. Epub 2007 Mar 23. PMID 17380255
- [Background] Whitlock RP, Crowther MA, Warkentin TE, Blackall MH, Farrokhyar F, Teoh KH. Warfarin cessation before cardiopulmonary bypass: lessons learned from a randomized controlled trial of oral vitamin K. Ann Thorac Surg. 2007 Jul;84(1):103-8. doi: 10.1016/j.athoracsur.2007.03.014. PMID 17588394
- [Background] Crowther MA, Ageno W, Schnurr T, Manfredi E, Kinnon K, Garcia D, Douketis JD. Oral vitamin K produces a normal INR within 24 hours of its administration in most patients discontinuing warfarin. Haematologica. 2005 Jan;90(1):137-9. PMID 15642685
- [Background] Ageno W, Garcia D, Silingardi M, Galli M, Crowther M. A randomized trial comparing 1 mg of oral vitamin K with no treatment in the management of warfarin-associated coagulopathy in patients with mechanical heart valves. J Am Coll Cardiol. 2005 Aug 16;46(4):732-3. doi: 10.1016/j.jacc.2005.05.022. No abstract available. PMID 16098445
- [Background] Wilson SE, Watson HG, Crowther MA. Low-dose oral vitamin K therapy for the management of asymptomatic patients with elevated international normalized ratios: a brief review. CMAJ. 2004 Mar 2;170(5):821-4. doi: 10.1503/cmaj.1030478. PMID 14993179
- [Background] Gunther KE, Conway G, Leibach L, Crowther MA. Low-dose oral vitamin K is safe and effective for outpatient management of patients with an INR>10. Thromb Res. 2004;113(3-4):205-9. doi: 10.1016/j.thromres.2004.03.004. PMID 15140584
- [Background] Crowther MA, Wilson S. Vitamin K for the treatment of asymptomatic coagulopathy associated with oral anticoagulant therapy. J Thromb Thrombolysis. 2003 Aug-Oct;16(1-2):69-72. doi: 10.1023/B:THRO.0000014597.87575.e9. PMID 14760216
- [Background] Ageno W, Crowther M, Steidl L, Ultori C, Mera V, Dentali F, Squizzato A, Marchesi C, Venco A. Low dose oral vitamin K to reverse acenocoumarol-induced coagulopathy: a randomized controlled trial. Thromb Haemost. 2002 Jul;88(1):48-51. PMID 12152676
- [Background] Crowther MA, McDonald E, Johnston M, Cook D. Vitamin K deficiency and D-dimer levels in the intensive care unit: a prospective cohort study. Blood Coagul Fibrinolysis. 2002 Jan;13(1):49-52. doi: 10.1097/00001721-200201000-00007. PMID 11994567
- [Background] Crowther MA, Julian J, McCarty D, Douketis J, Kovacs M, Biagoni L, Schnurr T, McGinnis J, Gent M, Hirsh J, Ginsberg J. Treatment of warfarin-associated coagulopathy with oral vitamin K: a randomised controlled trial. Lancet. 2000 Nov 4;356(9241):1551-3. doi: 10.1016/S0140-6736(00)03125-1. PMID 11075768
- [Background] Crowther MA, Donovan D, Harrison L, McGinnis J, Ginsberg J. Low-dose oral vitamin K reliably reverses over-anticoagulation due to warfarin. Thromb Haemost. 1998 Jun;79(6):1116-8. PMID 9657434
- [Background] Clark NP, Witt DM, Delate T, Trapp M, Garcia D, Ageno W, Hylek EM, Crowther MA; Warfarin-Associated Research Projects and Other Endeavors Consortium. Thromboembolic consequences of subtherapeutic anticoagulation in patients stabilized on warfarin therapy: the low INR study. Pharmacotherapy. 2008 Aug;28(8):960-7. doi: 10.1592/phco.28.8.960. PMID 18657012
- [Background] Carlquist JF, Horne BD, Muhlestein JB, Lappe DL, Whiting BM, Kolek MJ, Clarke JL, James BC, Anderson JL. Genotypes of the cytochrome p450 isoform, CYP2C9, and the vitamin K epoxide reductase complex subunit 1 conjointly determine stable warfarin dose: a prospective study. J Thromb Thrombolysis. 2006 Dec;22(3):191-7. doi: 10.1007/s11239-006-9030-7. PMID 17111199
- [Background] Schulman S, Beyth RJ, Kearon C, Levine MN. Hemorrhagic complications of anticoagulant and thrombolytic treatment: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):257S-298S. doi: 10.1378/chest.08-0674. PMID 18574268
- [Background] Proportion Difference Power / Sample Size Calculation. 8-7-2008.
- [Derived] Boonyawat K, Wang L, Lazo-Langner A, Kovacs MJ, Yeo E, Schnurr T, Schulman S, Crowther MA. The effect of low-dose oral vitamin K supplementation on INR stability in patients receiving warfarin. A randomised trial. Thromb Haemost. 2016 Aug 30;116(3):480-5. doi: 10.1160/TH16-04-0320. Epub 2016 Jun 23. PMID 27346552
- See also: A webinar describing results of our prior study may be found at this website — http://www.acforum.org/